CLINICAL TRIAL: NCT05831852
Title: Screening of the Possible Risk Factors for Borderline Personality Disorders Using Validated Arabic Version of Maclean Screening Tool: A Study in the Egyptian University Students "
Brief Title: Screening of the Possible Risk Factors for Borderline Personality Disorders and Validation of Maclean Instrument
Status: Completed | Type: Observational
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Sara ElAdawy, lecturer of clinical pharmacy, October University for Modern Sciences and Arts
Other Study IDs: RSPL 2.2
Record Dates: First submitted 2023-04-16; First posted 2023-04-26 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Borderline Personality Disorder
Keywords: BPD; Maclean instrument; validation; risk factors
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one group
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Borderline personality disorder is a mental illness that severely impacts a person's ability to regulate their emotions. This loss of emotional control can increase impulsivity, affect how a person feels about themselves, and negatively impact their relationships with others. In fact, the societal impact of BPDs might be found in emotional suffering, disability and economic burden. In addition in BPD, the suicide rate might be as high as 8-10%. the presence of BPD also interferes with response to treatment of physical and psychiatric comorbidities, such as migraine, HIV, anxiety disorders and substance use disorders. Furthermore, BPD in particular, are associated with high rates of unemployment, absences from work and inefficiency at work, with only 25% of patients suffering from BPD working full time and 40% receiving disability payments. Accordingly, early detection and management would be of great societal and economic impact. Our Study aim is to validate the Arabic version of Maclean Instrument for screening and detection of BPD and and investigate the possible risk factors associated with that disease

DETAILED DESCRIPTION:
Borderline personality disorder (BPD) is a mental health problem that affects the way you feel about yourself and others, the way you think , difficulty in managing behavior and emotions, self-image issues and a pattern of relationships that are unstable. BPD patients frequently describe their life as unpredictable and stressful. As stated in the Diagnostic and Statistical Manual of Mental Disorders (5th ed.), borderline personality disorder (BPD) is a serious mental illness characterized by a pervasive pattern of instability in interpersonal relationships, self-image and effect, as well as marked impulsivity. This condition arises in early adulthood or adolescence, leading to severe functional impairment and subjective discomfort. Unfortunately, diagnosis and treatment of BPD is often delayed, leading to a less favorable outcome. This is especially true in patients with early onset BPD, in whom the detection and subsequent therapeutic intervention on the disorder is usually further put off. Indeed, in the last two decades, there has been a great sensibilization towards personality disorder (PD)diagnosis in adolescence, reflected in the significant increase in empirical studies regarding this matter, and in the legitimization of adolescent PD diagnosis in psychiatric nomenclature (DSM-5 and ICD-11), as well as in national treatment guidelines in the UK and Australia. Nonetheless, a recent review by Sharp has stressed how scientific evidence and national practice guidelines are yet to penetrate routine clinical care. Indeed, in common clinical practice diagnosis and consequently, treatment of BPD is usually delayed due to underestimation of symptoms and, often, hesitation to diagnose this disorder in younger individuals. BPD is progressively considered a life expectancy formative disorder that exists on a layered continuum of severity. The recent studies for the adults who have BDP disease couldn't find a pharmacological treatment for them. The symptoms treatment with pharmacotherapy is not accurate for the treatment of BDP in adults, the pharmacotherapy should not be used for adolescent BPD. The only study exist is about the using of omega-3 fatty acids and the increase risk of psychosis. Overall, there is no pharmacological treatment for the BDP disease for adults, also the risks of iatrogenic and poly-pharmacy toxicity is high in these young people. The other comorbidities of the disease are treated from the clinical for adolescents, using the pharmacological therapy when needed. Our study aim is to validate the Arabic version of Maclean Instrument for screening and detection of BPD and and investigate the possible risk factors associated that disease thus decreasing the societal and economic burden of that disease

ELIGIBILITY:
Inclusion Criteria:

* age group (18-28 years old )
* University students

Exclusion Criteria:

* less than 18 years old
* more than 28 years old

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: adults
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
validation of Arabic version of Maclean Instrument | 6 months
  detection of reliability and consistency
Detection of Borderline personality disorder Risk factors in Egyptians students | 6 months
  survey

CONTACTS AND LOCATIONS:
Overall Officials: sara Eladawy, PhD, Principal Investigator — MSA university; mohamed hafez, Study Director — biostatistician, biomedical informatics medical research institute Alexandria University; mohamed emad, Study Chair — biostatistician, biomedical informatics, medical research institute, Alexandria University
Locations (1):
- October University for modern sciences and arts, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dias DS, Natividade JC. Brazilian adaptation of the McLean Screening Instrument for Borderline Personality Disorder. Trends Psychiatry Psychother. 2024;46:e20220486. doi: 10.47626/2237-6089-2022-0486. Epub 2022 Oct 18. PMID 36257605